CLINICAL TRIAL: NCT03433001
Title: A Prospective, Multicenter, Observational Study in Relapsed and/or Refractory Multiple Myeloma Patients Treated With Ixazomib Plus Lenalidomide and Dexamethasone
Brief Title: A Study in Relapsed and/or Refractory Multiple Myeloma Patients Treated With Ixazomib Plus Lenalidomide and Dexamethasone
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16042; JapicCTI-183860 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2022-05

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ixazomib + Lenalidomide + Dexamethasone: Participants took ixazomib, lenalidomide, and dexamethasone under conditions of standard medical care in this study. The dosage and administration of ixazomib, lenalidomide, and dexamethasone were not defined by the protocol but according to the package insert of each drug.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The purpose of this study is to investigate the real world effectiveness and safety of ixazomib in combination with lenalidomide and dexamethasone (IRd) in patients with relapsed and/or refractory multiple myeloma (RRMM), under conditions of standard medical care. In addition, an exploratory study of biomarkers will be conducted.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib. Ixazomib is being tested to treat people who have relapsed and/or refractory multiple myeloma (RRMM) under the conditions of standard medical care. This study is a non-interventional (observational), domestic, multicenter, prospective study in patients with RRMM. This study will look at the effectiveness and safety of ixazomib in combination with lenalidomide and dexamethasone in Japanese patients with RRMM as standard medical care. In addition, an exploratory study of biomarkers will be conducted in this study.

The study will enroll approximately 300 patients. All participants will receive Ixazomib + Lenalidomide + Dexamethasone (IRd) therapy as standard medical care.

This multi-center trial will be conducted in Japan. The overall time of observational period in this study will be 36 months. For each participant, the observation period will be from the start of IRd therapy until either 24 months after the enrollment date of the final patient to enroll, or until death or withdrawal of consent, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 20 years or older at the time of enrollment
2. Patients with RRMM
3. Participants who are scheduled to start IRd therapy
4. Participants who can provide written informed consent of their own free will before the start of study treatment
5. Participants who are judged by the principal investigator or investigator(s) to have the faculty to understand and comply with the requirements of the study

Exclusion Criteria:

1. Female Participants who are nursing or pregnant
2. Participants who have been treated with ixazomib
3. Participants with hypersensitivity to any of the components of IRd therapy, their analogs or excipients
4. Participants with another active malignancy, i.e. synchronous active malignancy or previous malignancy with a disease-free period of less than 5 years, except for participants with carcinoma in situ (intraepithelial carcinoma) or intramucosal carcinoma judged to be cured by topical treatment
5. Participants who are not registered with, or comply with, the guidelines of the lenalidomide management program
6. Participants who, in the judgement of the principal investigator or investigator(s), are considered to be unsuitable for enrolment into the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult men and women who have a confirmed diagnosis of multiple myeloma, who is scheduled to begin treatment with IRd due to relapsed and/or refractory disease, and who meet other eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kogure Y, Handa H, Ito Y, Ri M, Horigome Y, Iino M, Harazaki Y, Kobayashi T, Abe M, Ishida T, Ito S, Iwasaki H, Kuroda J, Shibayama H, Sunami K, Takamatsu H, Tamura H, Hayashi T, Akagi K, Shinozaki T, Yoshida T, Mori I, Iida S, Maeda T, Kataoka K. ctDNA improves prognostic prediction for patients with relapsed/refractory MM receiving ixazomib, lenalidomide, and dexamethasone. Blood. 2024 Jun 6;143(23):2401-2413. doi: 10.1182/blood.2023022540. PMID 38427753
- [Derived] Horigome Y, Iino M, Harazaki Y, Kobayashi T, Handa H, Hiramatsu Y, Kuroi T, Tanimoto K, Matsue K, Abe M, Ishida T, Ito S, Iwasaki H, Kuroda J, Shibayama H, Sunami K, Takamatsu H, Tamura H, Hayashi T, Akagi K, Maeda T, Yoshida T, Mori I, Shinozaki T, Iida S. A prospective, multicenter, observational study of ixazomib plus lenalidomide-dexamethasone in patients with relapsed/refractory multiple myeloma in Japan. Ann Hematol. 2024 Feb;103(2):475-488. doi: 10.1007/s00277-023-05428-7. Epub 2023 Sep 11. PMID 37695378
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60204db2bf003ab49576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant s took part in the survey at 101 investigative sites in Japan, from 2 April 2018 to 11 June 2021.
Pre-assignment Details: A total of 295 participants were enrolled and received the study treatment in this study.
Period: Overall Study
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Started | 295
Completed | 66
Not Completed | 229
Not completed — Lack of Efficacy | 109
Not completed — Adverse Event | 69
Not completed — Withdrawal by Subject | 10
Not completed — Death | 12
Not completed — Lost to Follow-up | 4
Not completed — Other | 25

BASELINE CHARACTERISTICS:
Population: Full Analysis Set, defined as all participants who were enrolled into the study and who receive at least one dose of ixazomib.
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 168
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 295
Hight [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 288
    (all) | 157.2 (9.70)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 277
    (all) | 56.91 (11.122)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2]] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2]
    number analyzed (Participants) | 276
    (all) | 22.96 (3.353)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Population: The number analyzed is the number of participants with data available for analysis.
  m^2
    number analyzed (Participants) | 276
    (all) | 1.562 (0.1830)
International Staging System (at Initial Diagnosis) [Count of Participants; unit: Participants] — International Staging System is a staging system for cancer progression. Stages are classified by Stage I to Stage III. Stage I: Serum beta2-microglobulin <3.5 mg/L and albumin ≥3.5 g/dL; Stage II: Neither Stage I or III, meaning that either: beta2-microglobulin level ≥3.5 and <5.5 mg/L (with any albumin level), OR albumin <3.5 g/dL with beta2-microglobulin <3.5 mg/L; Stage III: Serum beta2-microglobulin ≥5.5 mg/L. Normal serum beta2-microglobulin: <3.0 mg/L; normal albumin: 3.5-5.0 g/dL.
  Participants
    Stage I | 78
    Stage II | 112
    Stage III | 101
    Missing | 4
International Staging System (at First Treatment) [Count of Participants; unit: Participants]
  Stage I | 130
  Stage II | 78
  Stage III | 31
  Missing | 56
Eastern Cooperative Oncology Group performance status (ECOG P.S.) [Count of Participants; unit: Participants] — ECOG P.S. assess participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory ( greater than [>] 50 percent [%] of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead.
  Participants
    0 | 147
    1 | 90
    2 | 23
    3 | 18
    4 | 5
    Missing | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the period from the start of ixazomib, lenalidomide, dexamethasone (IRd) therapy in standard medical care to the time of confirmed progressive disease (PD) or confirmed death (regardless of the cause of death), whichever was earlier. PFS was assessed by International Myeloma Working Group (IMWG) Criteria (2014 version). Per IMWG criteria, PD: serum M-component increase ≥ 0.5 g/dl or urine M-component increase ≥ 200 mg/24-hour/ difference between involved and uninvolved free light chain (FLC) levels increase >10 mg/dl or bone marrow plasma cell ≥ 10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 36 Months as a maximum
Population: as for baseline characteristics
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Months | 4.79 (3.34)

2. Secondary Outcome: PFS Rate at 12 Months and 24 Months After the Start of Treatment
Description: PFS rate was defined as the percentage of participants who were alive and have not had disease progression at 12 months and 24 months after the date of start of study treatment. PFS was assessed by IMWG Criteria (2014 version). Per IMWG criteria, PD: serum M-component increase ≥ 0.5 g/dl or urine M-component increase ≥ 200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell ≥ 10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: 12 months and 24 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants
  Month 12 | 57 [51 to 63]
  Month 24 | 41 [35 to 47]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the period from the start of IRd therapy in standard medical care to the time when death (regardless of the cause of death) is confirmed.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Months | 20.23 (14.28)

4. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including partial response (PR), very good PR (VGPR) and complete response (CR) assessed with IMWG Criteria after each cycle of treatment. Per IMWG criteria, PR: ≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved free light chain (FLC) levels/ ≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/ ≥50% reduction in size of soft tissue plasmacytomas. VGPR: serum+urine M-protein detectable by immunofixation but not on electrophoresis/ ≥90% reduction in serum M-protein+urine M-protein level <100 mg/24-hour. CR: negative immunofixation on serum+urine +disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants
  CR | 20.0
  VGPR | 8.5
  PR | 22.0

5. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT will be measured as the period from the start of IRd therapy in standard medical care to the start of next treatment or time when death is confirmed (regardless of the cause of death), whichever is earlier.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Months | 5.02 (4.43)

6. Secondary Outcome: Duration of Therapy (DOT)
Description: DOT is defined as the treatment duration of IRd therapy.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Days | 353.3 (320.07)

7. Secondary Outcome: Percentage of Participants Who Continue to Receive Treatment at 12 Months and 24 Months After Start of Treatment
Time Frame: 12 months and 24 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants
  Month 12 | 40.0 [34.4 to 45.8]
  Month 24 | 21.7 [17.1 to 26.8]

8. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve a best response of PR or better including stringent complete response (sCR), VGPR and PR assessed with IMWG Criteria, after the start of the study treatment.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants | 53.9 [48.0 to 59.7]

9. Secondary Outcome: Percentage of Participants Who Achieve VGPR or Better (CR+VGPR)
Description: The percentage of participants of CR + VGPR is defined as the rate of participants who achieve a best response of VGPR or better (sCR, CR, or VGPR) according to the IMWG Criteria after the start of the IRd therapy.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants | 31.5 [26.3 to 37.2]

10. Secondary Outcome: Patient-Reported Outcome Health-Related Quality of Life (HRQoL) Based on European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Global Health Status Score
Description: EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale. EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores of Global Health Status in EORTC QLQ-C30 were linearly transformed to a total score between 0-100 and reported, with a high score indicating better QOL.
Time Frame: Baseline and End of Treatment (Up to 37 cycles, each cycle was of 28 days)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 279
Score on a Scale
  Baseline | 59.95 (22.472)
  End of Treatment: number analyzed (Participants) | 2
  End of Treatment | 75.00 (11.785)

11. Secondary Outcome: Patient-Reported Outcome HRQoL Based on EORTC Multiple Myeloma Module (EORTC QLQ-MY20) Score
Description: EORTC QLQ-MY20 has 20 items across 4 independent subscales, 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms, and side effects of treatment). Scores are averaged, and transformed to 0-100 scale. For the future perspective scale, higher score = better perspective of the future. For the body image scale, higher scores = better body image. Higher score for the disease symptoms scale = higher level of symptomatology.
Time Frame: Baseline and End of Treatment (Up to 37 cycles, each cycle was of 28 days)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 278
Score on a Scale
  Disease Symptoms: Baseline | 19.33 (18.949)
  Disease Symptoms: End of Treatment: number analyzed (Participants) | 2
  Disease Symptoms: End of Treatment | 11.11 (7.857)
  Side-Effects of Treatment: Baseline | 17.80 (13.903)
  Side-Effects of Treatment: End of Treatment: number analyzed (Participants) | 2
  Side-Effects of Treatment: End of Treatment | 16.67 (7.857)
  Body Image: Baseline | 28.18 (30.397)
  Body Image: End of Treatment: number analyzed (Participants) | 2
  Body Image: End of Treatment | 16.67 (23.570)
  Future Perspective: Baseline | 42.49 (25.634)
  Future Perspective: End of Treatment: number analyzed (Participants) | 2
  Future Perspective: End of Treatment | 33.33 (0.000)

12. Secondary Outcome: Rate of Minimal Residual Disease (MRD) Negativity in Bone Marrow in Participants Who Achieved CR
Description: Rate of MRD will be calculated by the percentage of participants who are MRD-negative.
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 68
Percentage of Participants
  10^-4=< - Max | 26.7
  10^-5=< - <10^-4 | 16.7
  10^-6=< - <10^-5 | 6.7
  Negative | 50.0

13. Secondary Outcome: Relative Dose Intensity (RDI)
Description: RDI is defined as 100*(Total amount of dose taken)/(Total prescribed dose of treated cycles), where total prescribed dose equals [dose prescribed at enrollment* number of prescribed doses per cycle* the number of treated cycles].
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percent
  Ixazomib | 66.49 (21.054)
  Lenalidomide | 44.72 (22.815)
  Dexamethasone | 41.07 (26.571)

14. Secondary Outcome: Percentage of Participants With Bone Lesions (Bone Evaluation)
Time Frame: Up to 36 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Percentage of Participants | 21.5 [12.3 to 33.5]

15. Secondary Outcome: Number of Participants Reporting One or More Treatment-Emergent AEs (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 36 months as a maximum
Population: Safety Analysis Set: all participants who were enrolled into the study and who receive at least one dose of any drug used in IRd therapy (i.e. ixazomib, lenalidomide, or dexamethasone)
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 295
Participants | 249

ADVERSE EVENTS:
Time Frame: Up to 36 months as a maximum
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib + Lenalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 24/295
Serious Adverse Events (participants affected / at risk) | 96/295
Other Adverse Events (participants affected / at risk) | 225/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib + Lenalidomide + Dexamethasone (N=295)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Colitis ischaemic (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Cardiac death (General disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 14
Cellulitis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Pneumonia influenzal (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 3
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar haemorrhage (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Renal disorder (Renal and urinary disorders) | 2
Nephropathy toxic (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib + Lenalidomide + Dexamethasone (N=295)
Anaemia (Blood and lymphatic system disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 72
Constipation (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 16
Malaise (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 16
Neutrophil count decreased (Investigations) | 76
Platelet count decreased (Investigations) | 75
White blood cell count decreased (Investigations) | 69
Rash (Skin and subcutaneous tissue disorders) | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03433001/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03433001/SAP_001.pdf